CLINICAL TRIAL: NCT06699511
Title: Effectiveness of Pilates in Patients With Subacute Low Back Pain
Acronym: Pilates-SLBP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, TUĞBA ŞAHBAZ, Assoc. Prof, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAEK/2022.11.211; KAEK/2022.11.211 (Other: Kanuni Sultan Suleyman Training and Research Hospital)
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Subacute Low Back Pain
Keywords: Pilates; Subacute low back pain
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study utilizes a parallel-group interventional study model to compare the effects of Pilates exercises versus a standard home exercise program on subacute low back pain. Participants are randomly assigned to one of two groups:
  Pilates Group: Participants in this group will receive a structured Pilates program targeting core stability, flexibility, and posture correction, which is specifically designed for low back pain management. Pilates exercises will be supervised by a qualified instructor to ensure proper technique and safety.
  Home Exercise Group: Participants in this group will follow a standard home exercise regimen tailored to relieve low back pain. These exercises focus on general strength and flexibility but are not specific to Pilates techniques.
  Both groups will participate in their respective programs for eight weeks. Outcomes, including pain levels, functional mobility, and quality of life, will be measured at three time points: baseline, post-treatment, and follow
Who Masked: Participant
Masking Description: In this clinical trial, masking will apply primarily to the Outcomes Assessor to ensure unbiased evaluation of results. The assessor, who will measure outcomes such as pain intensity, mobility, and quality of life, will be unaware of which intervention group (Pilates or home exercise) each participant belongs to. This masking minimizes the risk of bias in interpreting results based on prior knowledge of the intervention received by participants.
  If there are additional parties involved in data analysis or reporting who might influence the results, they will also be masked to the intervention assignments to maintain the integrity of the study outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pilates exercise (Active Comparator): pilates exercise
  Interventions: Behavioral: Exercise
- Home exercis (Active Comparator): Home exercise
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise

SUMMARY:
This study aims to evaluate the effectiveness of Pilates exercises in patients with subacute low back pain, which typically lasts between 4 and 12 weeks. Subacute low back pain is longer-lasting than acute pain and can negatively impact daily activities and quality of life. Pilates is an exercise method that strengthens core muscle groups, improves flexibility, and supports body balance.

This research is designed as a comparative study between two groups. One group will participate in Pilates exercises, while the other group will follow a standard home exercise program. The study will assess outcomes such as pain level, mobility, and quality of life. Through this, the study aims to provide more insights into the potential of Pilates as a treatment method for subacute low back pain.

DETAILED DESCRIPTION:
This study investigates the role of Pilates exercises in managing subacute low back pain, a condition defined as lasting between 4 and 12 weeks. Subacute low back pain often disrupts daily functioning and lowers quality of life, and effective interventions during this stage are crucial to prevent the transition to chronic pain. Pilates has been suggested as a beneficial exercise approach due to its focus on core stability, flexibility, and balanced body mechanics, which may reduce pain and improve functional outcomes in low back pain patients.

Participants in the study will be divided into two groups: a Pilates group and a home exercise group. The Pilates group will participate in a structured Pilates program designed to target core muscle strength and flexibility over a set period, while the home exercise group will follow a standard exercise program tailored for general low back pain relief. Both groups will perform their respective exercises for eight weeks.

The primary outcome measures will include pain intensity, physical function, and quality of life, assessed at baseline, post-treatment, and follow-up periods. The findings from this study will contribute to understanding whether Pilates can be a valuable addition to conservative treatment approaches for subacute low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 65 years.D
* Diagnosis of subacute low back pain, defined as pain lasting between 6 and 12 weeks
* No previous Pilates experience.

Exclusion Criteria:

* History of spinal surgery or significant spinal deformities (e.g., scoliosis).
* Presence of serious medical conditions such as cardiovascular disease, uncontrolled hypertension, or neurological disorders.
* Pregnancy or planned pregnancy during the study period.
* Use of pain-relief medications that could interfere with the results of the study.
* Participation in any structured physical therapy program in the last three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | pretreatment, post-treatment (8 weeks), and at 3-month follow-up
  The Visual Analog Scale (VAS) is used to measure pain intensity. The scale ranges from 0 to 10, where 0 represents 'no pain' and 10 represents 'worst possible pain.' Higher scores indicate worse outcomes, signifying greater pain intensity

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Beykent Univesity, Istanbul, Büyükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share IPD is currently under consideration and will depend on future funding resources and availability of data-sharing infrastructure.

REFERENCES:
- [Derived] Asik HK, Sahbaz T. Preventing chronic low back pain: investigating the role of Pilates in subacute management-a randomized controlled trial. Ir J Med Sci. 2025 Jun;194(3):949-956. doi: 10.1007/s11845-025-03939-y. Epub 2025 Apr 4. PMID 40183915
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34847915/
- Available data/document: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/34847915/